CLINICAL TRIAL: NCT01398358
Title: Enhancing Self Regulation as a Strategy for Obesity Prevention in Head Start Preschoolers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: Michigan State University (Other)
Responsible Party: Principal Investigator, Julie Lumeng, Associate Professor of Pediatrics, University of Michigan
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2010-04785
Record Dates: First submitted 2011-07-19; First posted 2011-07-20 (Estimated); Results first posted 2018-02-05 (Actual); Last update posted 2018-02-05 (Actual); Status verified 2017-07

CONDITIONS: Obesity
Keywords: obesity; prevention; children
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Usual Head Start Exposure (No Intervention): Children will attend their usual Head Start classroom and receive the usual educational interventions provided in that classroom.
- Parents of Preschoolers Series (POPS) (Experimental): Children attend Head Start preschool. Within the classroom, they receive a series of lessons about nutrition and obesity prevention delivered by an Extension Educator in collaboration with the classroom teacher. Parents are invited to attend a series of classes about nutrition and obesity prevention.
  Interventions: Behavioral: Parents of Preschoolers Series
- POPS + Incredible Years Series (IYS) (Experimental): Children attend Head Start preschool. Within the classroom, they receive a series of lessons about nutrition and obesity prevention delivered by an Extension Educator in collaboration with the classroom teacher. Parents are invited to attend a series of classes about nutrition and obesity prevention. In the classroom, children also receive a series of lessons about emotional and behavioral self-regulation delivered by a trained mental health specialist. The parents also are invited to classes about child behavioral and emotional self-regulation delivered by a mental health specialist.
  Interventions: Behavioral: Parents of Preschoolers Series; Behavioral: Incredible Years Series

INTERVENTIONS:
Behavioral: Parents of Preschoolers Series — The POPS-Parent intervention consists of eight 60-90 minute lessons about preventing childhood obesity followed by four 10-minute reinforcing telephone contacts. Each lesson includes opportunities for parents to develop and practice skills, and a discussion of strategies to overcome challenges and problem-solving techniques, with an emphasis on building knowledge and self-efficacy.
  The POPS-Child Intervention uses children's stories with embedded healthy nutrition themes. Five lessons (6 books) are delivered over 12 weeks. Activities include classroom cooking experiences, games/activities associated with the story's nutrition themes, and goal setting. "Family Links" and "Parent Pages" are sent home to reinforce content from school to home.
  Arms: POPS + Incredible Years Series (IYS); Parents of Preschoolers Series (POPS)
Behavioral: Incredible Years Series — The Parent component (BASIC) is a group-based program (12-14 weeks, 2 hours/week) focused on enhancing parenting skills such as using effective praise, incentives, and limit-setting, and handling misbehavior. Parents complete homework activities that will be reviewed in group sessions and receive follow-up reinforcement phone calls.
  For the Child component ("Dinosaur School"), 60, 15-20 minute lessons are delivered during "Circle Time" in Head Start classrooms followed by small group activities. The curriculum focuses on teaching self-regulation skills, problem-solving strategies, and prosocial behaviors.
  Teachers are trained in classroom management strategies.
  Arms: POPS + Incredible Years Series (IYS)

SUMMARY:
The goal of this integrated project targeting the Childhood Obesity Prevention Challenge Area is to reduce the prevalence of obesity among children attending Head Start in Michigan. The proposed intervention program is based on Social Cognitive theory and the premise that enhancing children's capacity for emotional and behavioral self-regulation is a key component of effective obesity prevention. A randomized controlled trial design is proposed to evaluate, among 600 Head Start children and their parents, the effectiveness of 2 approaches to obesity prevention: (1) the Parents of Preschoolers Prevention Series (POPS), a curriculum delivered to preschoolers and their parents focused on obesity-related health behaviors; and (2) POPS in combination with the Incredible Years Series (IYS), an evidence-based program designed to improve preschoolers' emotional and behavioral self-regulation. The research objective is to test the hypotheses that: (1) POPS, compared to Usual Head Start exposure, will lead to greater improvements in obesity-related health behaviors and adiposity indices; and (2) POPS + IYS will lead to the greatest improvements in obesity-related health behaviors and adiposity indices, and this effect will be mediated by improved self-regulation. The extension objective is to evaluate the feasibility, fidelity, and educational effectiveness of the POPS and POPS + IYS interventions, as delivered by paraprofessionals and educators within Extension and Head Start. The education objective is to provide Extension and Head Start staff non-formal training and educational curricula which can be widely disseminated. The long-term goal of this project is disseminate a novel and effective approach to obesity prevention in preschoolers.

ELIGIBILITY:
Inclusion Criteria:

* child is enrolled in Head Start

Exclusion Criteria:

* Significant developmental disabilities that would preclude participation
* Child is a foster child
* Parent is non-English speaking

Ages: 2 Years to 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 697 (Actual)
Dates: Start 2011-03; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Julie Lumeng, MD, Principal Investigator — University of Michigan
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States

REFERENCES:
- [Background] Miller AL, Horodynski MA, Herb HE, Peterson KE, Contreras D, Kaciroti N, Staples-Watson J, Lumeng JC. Enhancing self-regulation as a strategy for obesity prevention in Head Start preschoolers: the growing healthy study. BMC Public Health. 2012 Nov 30;12:1040. doi: 10.1186/1471-2458-12-1040. PMID 23194185
- [Derived] Jansen EC, Miller AL, Lumeng JC, Kaciroti N, Brophy Herb HE, Horodynski MA, Contreras D, Peterson KE. Externalizing behavior is prospectively associated with intake of added sugar and sodium among low socioeconomic status preschoolers in a sex-specific manner. Int J Behav Nutr Phys Act. 2017 Oct 3;14(1):135. doi: 10.1186/s12966-017-0591-y. PMID 28974224

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 1150 assessed for eligibility
Pre-assignment Details: 417 declined to enroll; 36 ineligible
Groups:
- Parents of Preschoolers Series (POPS): Children attend Head Start preschool. Within the classroom, they receive a series of lessons about nutrition and obesity prevention delivered by an Extension Educator in collaboration with the classroom teacher. Parents are invited to attend a series of classes about nutrition and obesity prevention.
  Parents of Preschoolers Series: The POPS-Parent intervention consists of eight 60-90 minute lessons about preventing childhood obesity followed by four 10-minute reinforcing telephone contacts. Each lesson includes opportunities for parents to develop and practice skills, and a discussion of strategies to overcome challenges and problem-solving techniques, with an emphasis on building knowledge and self-efficacy.
  The POPS-Child Intervention uses children's stories with embedded healthy nutrition themes. Five lessons (6 books) are delivered over 12 weeks. Activities include classroom cooking experiences, games/activities associated with the story's nutrition themes, and goal
- POPS + Incredible Years Series (IYS): Children attend Head Start preschool. Within the classroom, they receive a series of lessons about nutrition and obesity prevention delivered by an Extension Educator in collaboration with the classroom teacher. Parents are invited to attend a series of classes about nutrition and obesity prevention. In the classroom, children also receive a series of lessons about emotional and behavioral self-regulation delivered by a trained mental health specialist. The parents also are invited to classes about child behavioral and emotional self-regulation delivered by a mental health specialist
  Parents of Preschoolers Series: The POPS-Parent intervention consists of eight 60-90 minute lessons about preventing childhood obesity followed by four 10-minute reinforcing telephone contacts. Each lesson includes opportunities for parents to develop and practice skills, and a discussion of strategies to overcome challenges and problem-solving techniques, with an emphasis on building knowledge an
Period: Overall Study
Arm/Group | Usual Head Start Exposure | Parents of Preschoolers Series (POPS) | POPS + Incredible Years Series (IYS)
Started | 218 | 224 | 255
Completed | 203 | 201 | 234
Not Completed | 15 | 23 | 21
Not completed — Lost to Follow-up | 11 | 21 | 18
Not completed — Withdrawal by Subject | 3 | 2 | 2
Not completed — no longer eligible | 1 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- POPS + Incredible Years Series (IYS): Children attend Head Start preschool. Within the classroom, they receive a series of lessons about nutrition and obesity prevention delivered by an Extension Educator in collaboration with the classroom teacher. Parents are invited to attend a series of classes about nutrition and obesity prevention. In the classroom, children also receive a series of lessons about emotional and behavioral self-regulation delivered by a trained mental health specialist. The parents also are invited to classes about child behavioral and emotional self-regulation delivered by a mental health specialist.
  Parents of Preschoolers Series: The POPS-Parent intervention consists of eight 60-90 minute lessons about preventing childhood obesity followed by four 10-minute reinforcing telephone contacts. Each lesson includes opportunities for parents to develop and practice skills, and a discussion of strategies to overcome challenges and problem-solving techniques, with an emphasis on building knowledge an
- Total: Total of all reporting groups
Arm/Group | Usual Head Start Exposure | Parents of Preschoolers Series (POPS) | POPS + Incredible Years Series (IYS) | Total
Number analyzed (Participants) | 218 | 224 | 255 | 697
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 218 | 224 | 255 | 697
  Between 18 and 65 years | 0 | 0 | 0 | 0
  >=65 years | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 4.12 (0.53) | 4.10 (0.52) | 4.12 (0.52) | 4.10 (0.50)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 117 | 110 | 131 | 358
  Male | 101 | 114 | 124 | 339
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 28 | 31 | 25 | 84
  Not Hispanic or Latino | 189 | 192 | 227 | 608
  Unknown or Not Reported | 1 | 1 | 3 | 5
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 1 | 0 | 2
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 56 | 93 | 70 | 219
  White | 129 | 99 | 159 | 387
  More than one race | 27 | 25 | 19 | 71
  Unknown or Not Reported | 5 | 6 | 7 | 18
Region of Enrollment [Number; unit: participants]
  United States | 218 | 224 | 255 | 697
Body Mass Index Z-score (BMI z-score) [Mean (Standard Deviation); unit: z-score] | 0.57 (1.03) | 0.62 (1.20) | 0.64 (1.28) | 0.61 (1.17)

OUTCOME MEASURES:

1. Primary Outcome: Change in Body Mass Index Z-score
Description: Child BMI z-score was calculated from measure height and weight at enrollment and at the end of the study period
Time Frame: 9 months
Population: Seven of the 697 were excluded from analysis because they were missing both pre- and post- intervention BMI z-score. It was possible for a child to be included in the final analysis population even if they had not completed the follow-up portion of the study because the mixed model statistical method used could include their pre-intervention data.
Measure: Mean (Standard Error); unit: Z-Score
Arm/Group | Usual Head Start Exposure | Parents of Preschoolers Series (POPS) | POPS + Incredible Years Series (IYS)
Number analyzed (Participants) | 216 | 221 | 253
Z-Score | -0.01 (0.03) | 0.00 (0.03) | -0.04 (0.03)

2. Secondary Outcome: Change in Teacher-reported Self-regulation as Measured by the General Adaptation T-score From the Social Competence and Behavior Evaluation Scale
Description: To assess self-regulation, teachers completed a modified 60-item version of the Social Competence and Behavior Evaluation (SCBE) scale.The SCBE assesses emotional and behavioral regulation difficulties typically seen in the preschool setting. It includes both positive (competence) and negative (emotional or behavioral problems) items, including internalizing (ie, anxious, sad) and externalizing (ie, oppositional) behaviors, both of which are indicators of poor behavioral self-regulation. The General Adaptation T-score assesses child overall emotional and behavioral self-regulation in the classroom setting. It is calculated by taking the mean of all 60 items for the SCBE questionnaire (with reverse scoring for questions capturing problem behavior) and then determining the corresponding t-score based on published tables. Higher scores indicate better self-regulation. The range for General Adaptation T-score is 30-70.
Time Frame: 9 months
Measure: Mean (Standard Error); unit: change in t-score from pre to post
Arm/Group | Usual Head Start Exposure | Parents of Preschoolers Series (POPS) | POPS + Incredible Years Series (IYS)
Number analyzed (Participants) | 216 | 221 | 253
change in t-score from pre to post | 0.93 (0.55) | 1.28 (0.56) | 3.92 (0.50)

ADVERSE EVENTS:
Time Frame: 9 months
Arm/Group | Usual Head Start Exposure | Parents of Preschoolers Series (POPS) | POPS + Incredible Years Series (IYS)
All-Cause Mortality (participants affected / at risk) | 0/218 | 0/224 | 0/255
Serious Adverse Events (participants affected / at risk) | 0/218 | 0/224 | 0/255
Other Adverse Events (participants affected / at risk) | 0/218 | 0/224 | 0/255

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes